CLINICAL TRIAL: NCT05410561
Title: Harnessing Telemedicine to Improve Alcohol Use Disorder Outcomes in Primary Care Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Allison Lin, Assistant Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00204315; 1R01AA029400-01 (NIH)
Record Dates: First submitted 2022-05-24; First posted 2022-06-08 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-06

CONDITIONS: Substance Use Disorders; Substance Use; Substance Dependence
Keywords: Telehealth; Cognitive behavioral therapy; Psychoeducation; Motivational interviewing; Alcohol consumption
MeSH Terms: conditions — Substance-Related Disorders; Alcohol Drinking

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TeleTx intervention (Experimental): The evidence-based manualized psychosocial program is via telehealth and uses adaptations of cognitive behavioral therapy and motivational interviewing.
  Interventions: Behavioral: TeleTx intervention
- Enhanced Usual Care (EUC) (Active Comparator): EUC will include brief psychoeducation about AUD and resources for treatment.
  Interventions: Behavioral: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: Enhanced Usual Care (EUC) — EUC will comprise one session of brief psychoeducation and referral information to alcohol use disorder (AUD) treatment.
  Arms: Enhanced Usual Care (EUC)
Behavioral: TeleTx intervention — TeleTx will consist of an initial session and then 8 ~counseling sessions.
  Arms: TeleTx intervention

SUMMARY:
The purpose of this trial is to test new programs to see if they might help people manage their health and health behaviors related to alcohol use and well-being. The program sessions focus on getting to know what's important to the participants, reviewing or setting goals, and using different skills and behaviors to better manage health. The trial will help the study team learn about ways to deliver health information in a way that is useful and interesting.

This research will take place remotely (e.g., Zoom, Facetime, Phone) and participants will be randomized to the Telehealth (TeleTx) group intervention or the Enhanced Usual Care (EUC) control group. Both groups will be asked to have follow-up visits up to 12 months from the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Current Diagnostic and Statistical Manual (DSM) -5 alcohol use disorder (AUD) based on alcohol symptom checklist
* An average of 3 or more drinking days per week for the past 30 days
* Have regular access to a device with video capabilities or a phone to use for study related calls

Exclusion Criteria:

* Inability to speak or understand English
* Conditions that preclude informed consent or understanding of assessment or intervention content
* Past 90-day AUD psychotherapy treatment,
* At elevated risk for complicated alcohol withdrawal
* Past-year drug injection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Alcohol Use Disorder Treatment Initiation | 3 months
  Percent of patients who initiate Alcohol Use Disorder psychotherapy treatment
Alcohol Use Disorder Treatment Engagement | 3 months
  Percent of patients who attend at least 2 additional Alcohol Use Disorder psychotherapy sessions
Alcohol consumption days | 3-months
  Percent days of alcohol use on the Timeline Follow Back interview
Alcohol consumption days | 6-months
  Percent days of alcohol use on the Timeline Follow Back interview
Alcohol consumption days | 12-months
  Percent days of alcohol use on the Timeline Follow Back interview
Heavy drinking days | 3-months
  Percent days heavy drinking on the Timeline Follow Back interview
Heavy drinking days | 6-months
  Percent days heavy drinking on the Timeline Follow Back interview
Heavy drinking days | 12-months
  Percent days heavy drinking on the Timeline Follow Back interview

SECONDARY OUTCOMES:
Total Alcohol Use Disorder Psychotherapy Treatment Attendance | 6-months
  Total number of psychotherapy sessions
Total Alcohol Use Disorder Psychotherapy Treatment Attendance | 12-months
  Total number of psychotherapy sessions
Drinking Risk Levels (Based on World Health Organization Cut-Offs) | Baseline to 3-months
  Change in WHO drinking levels (defined by alcohol consumed per day from 1g to undefined maximum with higher amounts associated with worse outcomes)
Drinking Risk Levels (Based on World Health Organization Cut-Offs) | Baseline to 6-months
  Change in WHO drinking levels (defined by alcohol consumed per day from 1g to undefined maximum with higher amounts associated with worse outcomes)
Drinking Risk Levels (Based on World Health Organization Cut-Offs) | Baseline to 12-months
  Change in WHO drinking levels (defined by alcohol consumed per day from 1g to undefined maximum with higher amounts associated with worse outcomes)
World Health Organization Quality of Life Abbreviated (WHO-QOL-BREF) | Baseline to 3-months
  Change in Quality of Life measure (WHO-QOL BREF). Transformed domain scores from 0 to 100. Higher scores denote better quality of life.
World Health Organization Quality of Life Abbreviated (WHO-QOL-BREF) | Baseline to 6-months
  Change in Quality of Life measure (WHO-QOL BREF). Transformed domain scores from 0 to 100. Higher scores denote better quality of life.
World Health Organization Quality of Life Abbreviated (WHO-QOL-BREF) | Baseline to 12-months
  Change in Quality of Life measure (WHO-QOL BREF). Transformed domain scores from 0 to 100. Higher scores denote better quality of life.
Alcohol consequences | Baseline to 3-months
  Change in alcohol consequences measured by the modified 17-item Short Inventory of Problem-R
Alcohol consequences | Baseline to 6-months
  Change in alcohol consequences measured by the modified 17-item Short Inventory of Problem-R
Alcohol consequences | Baseline to 12-months
  Change in alcohol consequences measured by the modified 17-item Short Inventory of Problem-R

CONTACTS AND LOCATIONS:
Overall Officials: Allison Lin, MD, Principal Investigator — University of Michigan; Erin Bonar, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - VA Ann Arbor Health Care | Veterans Affairs, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bonar EE, Goldstick JE, Rostker MJ, Dailey SE, Augustiniak AN, Brin C, Manderachia DA, Bourque C, Girard R, Sulkowski L, Lin LA. Testing a new model of telehealth-delivered treatment for primary care patients with alcohol use disorder: A randomized controlled trial protocol. Contemp Clin Trials. 2024 Jul;142:107549. doi: 10.1016/j.cct.2024.107549. Epub 2024 Apr 26. PMID 38679140